CLINICAL TRIAL: NCT00022204
Title: Double-Blind, Placebo-Controlled, Randomised Trial Of Alpha-Tocopherol And Oxpentifylline In Patients With Radiation Fibrosis
Brief Title: Vitamin E and Pentoxifylline in Treating Women With Lymphedema After Radiation Therapy for Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: CDR0000068794; RM-1597; EU-20050
Record Dates: First submitted 2001-08-10; First posted 2004-02-04 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2007-05

CONDITIONS: Breast Cancer; Lymphedema
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; lymphedema; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Lymphedema; Breast Neoplasms, Male | interventions — Vitamin E; Pentoxifylline

INTERVENTIONS:
Dietary Supplement: vitamin E
Drug: pentoxifylline
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Vitamin E and pentoxifylline may be effective in decreasing lymphedema in women who have received radiation therapy for breast cancer.

PURPOSE: Randomized phase II trial to determine the effectiveness of combining vitamin E and pentoxifylline in treating women who have lymphedema after receiving radiation therapy for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effects of vitamin E and pentoxifylline on lymphedema in patients previously treated with radiotherapy for breast cancer. II. Compare the normal tissue injury and quality of life in patients treated with this regimen vs placebo.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are randomized to one of two treatment arms. Arm I: Patients receive oral vitamin E and oral pentoxifylline twice daily for 6 months. Arm II: Patients receive oral placebo twice daily for 6 months. Quality of life is assessed at baseline and at 3, 6, 9, and 12 months. Patients are followed at 6 and 12 months.

PROJECTED ACCRUAL: A total of 100 patients (50 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Prior diagnosis of breast cancer T1-3, N0-1, M0 Prior radiotherapy to breast/chest wall plus axilla and/or supraclavicular fossa At least 2 years since prior radiotherapy No disease recurrence Arm lymphedema due to prior radiotherapy Reduced shoulder movement, induration in breast/chest wall, radiation-induced brachial plexopathy, symptomatic lung fibrosis, or non-healing wounds (including fractures) allowed as evidence of disability in addition to arm lymphedema Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: Not specified Sex: Female or male Menopausal status: Not specified Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: No liver failure Renal: No renal failure Cardiovascular: No ischemic heart disease No hypertension No hypotension No acute myocardial infarction No prior cerebral hemorrhage No prior retinal hemorrhage Other: Not pregnant Negative pregnancy test Fertile patients must use effective contraception No allergy to coconut oil

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: No concurrent insulin Radiotherapy: See Disease Characteristics Surgery: No prior axillary surgery Lower axillary sampling allowed Other: At least 3 months since prior daily vitamin E supplementation of more than 30 mg/day No prior pentoxifylline after radiotherapy No concurrent ketorolac or vitamin K No other concurrent vitamin E supplementation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-01

CONTACTS AND LOCATIONS:
Overall Officials: John R. Yarnold, MD, FRCR, Study Chair — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital, Sutton, England, United Kingdom

REFERENCES:
- [Result] Gothard L, Cornes P, Earl J, Hall E, MacLaren J, Mortimer P, Peacock J, Peckitt C, Woods M, Yarnold J. Double-blind placebo-controlled randomised trial of vitamin E and pentoxifylline in patients with chronic arm lymphoedema and fibrosis after surgery and radiotherapy for breast cancer. Radiother Oncol. 2004 Nov;73(2):133-9. doi: 10.1016/j.radonc.2004.09.013. PMID 15542159